CLINICAL TRIAL: NCT05250791
Title: A Randomised Feasibility Study Evaluating the Effect of Perioperative Intravenous Lidocaine on Colorectal Cancer Outcome After Surgery
Brief Title: Feasibility Study of Lidocaine Infusion During Bowel Cancer Surgery for Cancer Outcome
Acronym: FLICOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21CX7298; 2021-006185-20 (EudraCT Number); NIHR301741 (Other Grant/Funding Number: National Institute for Health Research); 1004491 (Registry Identifier: IRAS number)
Record Dates: First submitted 2022-01-28; First posted 2022-02-22 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer; Quality of Life; Recurrent Cancer
Keywords: Perioperative; Intravenous lidocaine; cancer recurrence; colorectal cancer; quality of life
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence | interventions — Lidocaine; Injections; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine (Active Comparator): An intravenous bolus of 2% lidocaine will be administered following the induction of anaesthesia at 1.5mg/kg ideal body weight over 20 minutes followed by intravenous infusion of 1.5 mg/kg/hour ideal body weight with a maximum rate of 120mg/hour for 24 hours.
  Interventions: Drug: Lidocaine hydrochloride 2% for injection
- 0.9% sterile Sodium Chloride solution for injection (Placebo Comparator): An equivalent infusion rate (ml) of placebo will be administered following the induction of anaesthesia over 20 minutes followed by hourly equivalent intravenous infusion in ml/hr of placebo with a maximum rate of 6mls/hr (equivalent of 120mg/hour for lidocaine) for 24 hours.
  Interventions: Drug: 0.9% sterile Sodium Chloride solution for injection

INTERVENTIONS:
Drug: Lidocaine hydrochloride 2% for injection — An intravenous bolus of 2% lidocaine will be administered following the induction of anaesthesia at 1.5mg/kg ideal body weight over 20 minutes followed by intravenous infusion of 1.5 mg/kg/hour ideal body weight with a maximum rate of 120mg/hour for 24 hours.
  Other Names: Xylocaine
  Arms: lidocaine
Drug: 0.9% sterile Sodium Chloride solution for injection — Administered as lidocaine
  Other Names: Saline
  Arms: 0.9% sterile Sodium Chloride solution for injection

SUMMARY:
This feasibility (small) study aims to see if it is possible to run a large study looking at the effect of lidocaine on large bowel cancer recurrence after surgery in the NHS hospitals.

DETAILED DESCRIPTION:
Strong preclinical evidence suggests that lidocaine, a type of local anaesthetic commonly used, could potentially reduce cancer recurrence if given during cancer surgery. This study will evaluate the feasibility of conducting a study comparing intravenous lidocaine infusion versus placebo administration for 24 hours from the start of general anaesthesia. The specific population will be any stage 2 or 3 colon or rectal cancer patient undergoing elective laparoscopic colorectal cancer surgery to look at postoperative cancer outcomes in two NHS settings. This study will explore the acceptability, facilitators and potential barriers of recruiting cancer patients, with possible anxieties of a new cancer diagnosis about to have major surgery along with other potential feasibility issues. It will also assess if follow-up and outcome data collection can be streamlined with usual care processes as much as possible and to guide the future definitive trial.

The project will:

1. Perform a feasibility study. This will be similar in design to the future bigger study and will see:

   * if there are any problems in giving lidocaine;
   * if patients and clinicians would be happy to take part in a study using a design where some patients get the drug and others get a non-active substance (known as placebo);
   * how many patients can we get from the different types and stages of bowel cancer;
   * if patients can be followed up successfully;
   * if we can collect all the data that we would need;
   * what measures might work well for the future study;
2. Look to see if blood tests can give some idea on how lidocaine might work in patients and if it can be confirmed in the bigger study.

The study will involve a small number of patients getting either lidocaine or placebo, and:

* filling in questionnaires to measure quality of life;
* follow up phone call at 6 and 12 months after surgery;
* having their records looked at to see if cancer comes back;
* both patients and clinicians to fill in a feedback questionnaire to see how they get on with the study processes;
* having extra blood tests before and after they finish the lidocaine/placebo infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above, undergoing laparoscopic surgery with stage 2 or 3 colon cancer
* Age 18 and above, undergoing laparoscopic surgery with stage 2 or 3 rectal cancer
* Ability and willingness to consent

Exclusion Criteria:

* Stage 1 and stage 4 colon or rectal cancer
* Palliative surgery with no curative intent
* Extensive comorbidities, i.e. American Society of Anesthesiologists (ASA) Score IV
* Patients with known or suspected allergy to lidocaine
* Patients who are currently pregnant* or breastfeeding
* Patients who are likely to have adverse effects from the accumulation of intravenous lidocaine:

  * current liver disease with a liver function outside the normal laboratory range
  * current renal failure (eGFR <30)
  * epilepsy
  * cardiac conduction abnormalities based on history and confirmed by electrocardiogram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | Baseline
  The number of eligible patients and the actual number recruited for colon and rectal cancer with stage 2 or 3.
Trial retention | 12 months post randomisation
  The number of participants who consent to participate who remain in the study until the end of follow up at 12 months.
The completion of data collection instruments | 6 months post randomisation
  on eCRF
The completion of data collection instruments | 12 months post randomisation
  on eCRF
Participant's feedback of study experiences | Day 3 hospital stay
  10 questions close-ended questionnaire with optional free text relating to informed consent procedures, the information given, the recruitment process and any suggestions for improvement.
Clinical staff feedback of study experiences | Day 3 hospital stay
  10 questions close-ended questionnaire with optional free text relating to informed consent procedures, the information given, the recruitment process and any suggestions for improvement.
Patients' reasons to refuse consent. | Baseline
  Patients who refuse consent will be asked for their reasons at the point of recruitment only
Clinicians' reasons for not recruiting patients. | Screening
  Clinicians will be asked their reasons for not recruiting patients

SECONDARY OUTCOMES:
Disease-free survival | 12-months post randomisation
  Cancer recurrence and death from any cause
Completion of EQ-5D-5L | Baseline
  The completeness of responses to the health-related quality of life questionnaire, EQ- 5D-5L which would be the outcome measure used in an economic evaluation as part of the definitive trial.
Completion of EQ-5D-5L | 6 months post randomisation
  The completeness of responses to the health-related quality of life questionnaire, EQ- 5D-5L which would be the outcome measure used in an economic evaluation as part of the definitive trial.
Completion of EQ-5D-5L | 12-months post randomisation
  The completeness of responses to the health-related quality of life questionnaire, EQ- 5D-5L which would be the outcome measure used in an economic evaluation as part of the definitive trial.
Completion of the cancer-specific quality of life questionnaires | Baseline
  Feasibility and completion of the Cancer-specific quality of life measured using the Functional Assessment of Cancer Therapy-Colorectal cancer (FACT-C) questionnaire.
Completion of the cancer-specific quality of life questionnaires | 6 months post randomisation
  Feasibility and completion of the Cancer-specific quality of life measured using the Functional Assessment of Cancer Therapy-Colorectal cancer (FACT-C) questionnaire.
Completion of the cancer-specific quality of life questionnaires | 12-months post randomisation
  Feasibility and completion of the Cancer-specific quality of life measured using the Functional Assessment of Cancer Therapy-Colorectal cancer (FACT-C) questionnaire.
Completion of healthcare and social care resource use questionnaires | 6 months post randomisation
  This will be a bespoke patient questionnaire on primary and secondary healthcare and social care resource use.
Completion of healthcare and social care resource use questionnaires | 12-months post randomisation
  This will be a bespoke patient questionnaire on primary and secondary healthcare and social care resource use.
Total hospital stays including readmission | 12-months post randomisation
  Recorded from medical notes and healthcare resource use form.

OTHER OUTCOMES:
Quantity of circulating free DNA | Day 3 hospital stay
  Change from baseline quantity of circulating free DNA at treatment completion
DNA whole-genome sequencing | Day 3 hospital stay
  Quantitative genomic analysis of the blood cells to study the characteristics and investigate the technical feasibility of this for the future definitive trial.
Quantity of circulating tumour cells | Day 3 hospital stay
  Change from baseline circulating tumour cells quantity at treatment completion
Circulating tumour cells functional characteristics | Day 3 hospital stay
  Comparison between lidocaine and placebo treatment group
Pro-inflammatory cytokine levels | Day 3 hospital stay
  Change from baseline pro-inflammatory cytokine levels at treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: West Raha, MBChB, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] West R, Soo CP, Murphy J, Vizcaychipi MP, Ma D. A protocol for a pilot study to assess the feasibility of a randomised clinical trial of perioperative intravenous lidocaine on colorectal cancer outcome after surgery (FLICOR trial). BJA Open. 2023 Jun;6:100138. doi: 10.1016/j.bjao.2023.100138. PMID 37387798